CLINICAL TRIAL: NCT06061718
Title: Multicenter, Open-label, Single-arm Trial to Evaluate the Safety and Efficacy of iDose® TR (Travoprost Intraocular Implant) in Conjunction With Cataract Surgery
Brief Title: Travoprost Intraocular Implant in Conjunction With Cataract Surgery
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLK-101-02
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- iDose TR (Experimental): Travoprost Intraocular Implant administered intracamerally in the study eye at the Day 1 Visit following successful cataract surgery
  Interventions: Drug: iDose TR

INTERVENTIONS:
Drug: iDose TR — anchored intracameral implant containing travoprost
  Other Names: travoprost intraocular implant

SUMMARY:
Subjects with cataract requiring extraction and who have open-angle glaucoma or ocular hypertension will undergo screening and washout from IOP-lowering medication, if applicable. Eligible subjects who meet all inclusion criteria and none of the exclusion criteria and who undergo successful cataract extraction with implantation of a posterior chamber intraocular lens (PC-IOL) will receive a travoprost intraocular implant and followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* clinically significant age-related cataract eligible for phacoemulsification in the study eye
* open-angle glaucoma or ocular hypertension in the study eye
* successful, uncomplicated cataract surgery using small incision phacoemulsification cataract surgery and insertion of a foldable posterior chamber IOL

Exclusion Criteria:

* unmedicated (washed out) IOP of >36 mmHg in the study eye
* hypersensitivity to travoprost or any other components of the travoprost intraocular implant
* vertical cup/disc ratio > 0.8 in the study eye
* best spectacle corrected visual acuity of worse than 20/80 in the fellow eye
* any ocular disease or condition that, in the opinion of the investigator, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean diurnal IOP | 3 months
  Mean diurnal IOP at the Month 3 Visit minus the mean diurnal IOP at the Baseline Visit

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Glaukos Corporation
Locations (1):
- Glaukos Clinical Study Site, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh IP, Voskanyan LA, Barber KM, Burden JH, Connolly L, Katz LJ, Usner DW, Kothe AC, Navratil T. Safety and efficacy of travoprost intracameral implant administered in combination with cataract surgery. Ther Adv Ophthalmol. 2025 Feb 14;17:25158414241310275. doi: 10.1177/25158414241310275. eCollection 2025 Jan-Dec. PMID 39959854